CLINICAL TRIAL: NCT05431491
Title: Feasibility of Slow Continuous Ultrafiltration With Regional Anticoagulation for Deresuscitation in Critically Ill Patients Though Standard Central or Peripheral Venous Access.
Brief Title: Feasibility of Slow Continuous UltraFiltration For Deresuscitation in Critically Ill Patients
Acronym: SCUFFD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Belfast Health and Social Care Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21021JS-AS
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2024-09

CONDITIONS: Fluid Overload
Keywords: Ultrafiltration; Deresuscitation
MeSH Terms: conditions — Edema | interventions — Ultrafiltration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ultrafiltration cohort (Experimental): These patients will be recruited into the study to assess the feasibility of slow continuous ultrafiltration through either a standard central venous catheter, or peripheral intravenous cannula.
  Interventions: Device: Ultrafiltration

INTERVENTIONS:
Device: Ultrafiltration — Ultrafiltration through much smaller intravenous cannula than what has previously been used.

SUMMARY:
To determine the feasibility and safety of deresuscitation using slow continuous ultrafiltration with regional citrate anticoagulation and peripheral or standard central venous access.

DETAILED DESCRIPTION:
Fluid deresuscitation has been shown to have favourable outcomes in the management of the critically ill patient. Whilst diuretic medications have previously been the mainstay of achieving this deresuscitation, the metabolic and biochemical complications associated with their use can limit their application. Mechanical ultrafiltration is another means of achieving fluid deresuscitation and has theoretical benefits over the use of intravenous diuretics. It allows a more titratable process, without the potential metabolic complications. The use of ultrafiltration has been limited by the requirement of wide bore central venous access. The SCUFFD study is a means of assessing whether ultrafiltration with regional anticoagulation can be achieved through standard central or peripheral venous access.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years)
* Evidence of fluid overload (greater than trace amount of peripheral oedema in >1 site, pulmonary oedema on chest radiograph, or positive fluid balance equivalent to >5% body weight)
* Clinician intention to target a negative fluid balance
* Expected to remain in a critical care setting beyond the next calendar day

Exclusion Criteria:

Anticipated unavailability of suitable vascular access

* Lack of commitment to full support
* Receiving or imminently planned to receive renal replacement therapy
* Hyponatraemia (Sodium <130mmol/L)
* Hypernatraemia (Sodium >150mmol/L)
* Significant metabolic alkalosis (Bicarbonate>30 and pH>7.5)
* Significant metabolic acidosis (HCO3- <18 mmol/l and pH < 7.30)
* Uncorrected hypokalaemia (Potassium <3.0mmol/L)
* Liver failure (Child-Pugh Grade B or above)
* Shock (any of: lactate >3mmol/L, extensive skin mottling, central capillary refill time>3 seconds, more than 1 vasoactive agent in use, noradrenaline dose >0.2 mcg/kg/min, use of dobutamine, adrenaline, milrinone, enoximone or levosimendan)
* Receiving any systemic anticoagulation other than for routine venous thromboembolism prophylaxis, or dual antiplatelet therapy
* Prisoner
* Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with daily fluid balance within 500 mL of prescribed target | 5 days per patient
  Assessing the feasibility of managing to achieve the target fluid balance
Number of patients with filter or circuit thrombosis requiring discontinuation of therapy | 5 days per patient
  Ensuring that the process of haemofiltration does not result in unacceptable levels of thrombotic events
Total volume of fluid removed using ultrafiltration | 5 days per patient
  Assessing the feasibility of fluid removal by ultrafiltration
Circuit lifespan | 5 days per patient
  The lifespan of each ultrafiltration circuit, to assess the feasibility of using this method as a therapeutic option

SECONDARY OUTCOMES:
Number of patients developing citrate accumulation | 5 days
  Defined as systemic total:ionised calcium ratio greater than 2.5
Number of patients developing metabolic alkalosis | 5 days
  Defined as new onset Bicarbonate>30 and pH >7.5
Number of patients developing metabolic acidosis | 5 days
  Defined as new onset Bicarbonate<18 and pH<7.30
Number of patients with a significant change in sodium | 5 days per patient
  Defined as new onset change in sodium >8mmol/l in 24 hours or less
Number of patients developing new onset hyponatraemia | 5 days per patient
  Defined as new onset sodium <130mmol/l
Number of patients developing new onset hypernatraemia | 5 days per patient
  Defined as new onset sodium >150mmol/l
Number of patients developing new onset hypokalaemia | 5 days per patient
  Defined as new onset potassium < 3mmol/l

CONTACTS AND LOCATIONS:
Overall Officials: Jon Silversides, PhD, Principal Investigator — BHSCT
Locations (1):
- Belfast City Hospital, Belfast, Down, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No personalized IPD will be available to be share with other researchers. Anonymised data will be grouped into a database which may be shared with other researchers.